CLINICAL TRIAL: NCT00240305
Title: A Randomised, Double-Blind, Placebo Controlled, Crossover Dose-Ranging Study to Investigate the Effect of Rosuvastatin (CRESTOR®) on High Density Lipoprotein Kinetics in Patients With the Metabolic Syndrome
Brief Title: A Study to Investigate the Effect of Rosuvastatin (CRESTOR®) on High Density Lipoprotein Kinetics in Patients With the Metabolic Syndrome
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 4522AS/0004
Record Dates: First submitted 2005-10-16; First posted 2005-10-18 (Estimated); Last update posted 2009-03-16 (Estimated); Status verified 2009-03

CONDITIONS: Metabolic Syndrome; Dyslipidemia
Keywords: Metabolic Syndrome; Dyslipidaemia
MeSH Terms: conditions — Metabolic Syndrome; Dyslipidemias | interventions — Rosuvastatin Calcium

INTERVENTIONS:
Drug: Rosuvastatin

SUMMARY:
The purpose of this study is to investigate the dose-related effect of treatment with rosuvastatin on production and fractional catabolism of apolipoprotein A-I (apoA-I) and apolipoprotein A-II (apoA-II), and on the plasma apoA-I, apoA-II and high-density lipoprotein cholesterol (HDL-C) concentration.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* male aged 30 to 70 years of age
* LDL-C <6 mmol/L
* HDL-C ≤1.2 mmol/L
* at least 2 of the following:
* insulin resistance (fasting glucose >6 mmol/L or insulin >10 mU/L or HOMA score >2.5)
* central obesity (waist circumference >=94 cm).
* plasma triglycerides >=1.7 and <4.5 mmol/L.
* blood pressure >=130/ >=85 mm Hg or on drug treatment for hypertension

Exclusion Criteria:

* LDL cholesterol >=6 mmol/L
* pre-existing or history of cardiovascular disease, diabetes, renal dysfunction, anaemia, history of significant dyspepsia or gastrointestinal disease
* apolipoprotein genotype E2/E2

Ages: 30 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15
Dates: Start 2004-04; Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
Determine the dose-related effect of treatment with rosuvastatin on production & fractional catabolism of apolipoprotein A-I (apoA-I) and apolipoprotein A-II (apoA-II), & on the plasma apoA-I, apoA-II & high-density lipoprotein cholesterol (HDL-C) c

SECONDARY OUTCOMES:
Determine the dose-related effect of treatment with rosuvastatin on cellular cholesterol efflux,total cholesterol, low-density lipoprotein cholesterol (LDL-C), non-LDL-C, triglyceride & pre1-HDL concentrations,HDL2,HDL3 cholesterol ratio
Cholesteryl ester transfer protein (CETP) and lecithin:cholesterol acyl transferase (LCAT) activity
Lathosterol and campesterol, total apolipoprotein B (apoB), nonesterified fatty acids (NEFA) and apolipoprotein C-III (apoC-III) plasma concentrations.

CONTACTS AND LOCATIONS:
Overall Officials: Gerald F. Watts, BSc PhD MD, Principal Investigator — University Department of Medicine, Royal Perth Hospital, University of Western Australia
Locations (1):
- Research Site, Perth, Western Australia, Australia

REFERENCES:
- [Derived] Ng TW, Ooi EM, Watts GF, Chan DC, Meikle PJ, Barrett PH. Association of Plasma Ceramides and Sphingomyelin With VLDL apoB-100 Fractional Catabolic Rate Before and After Rosuvastatin Treatment. J Clin Endocrinol Metab. 2015 Jun;100(6):2497-501. doi: 10.1210/jc.2014-4348. Epub 2015 Mar 27. PMID 25816050
- [Derived] Ng TW, Ooi EM, Watts GF, Chan DC, Weir JM, Meikle PJ, Barrett PH. Dose-dependent effects of rosuvastatin on the plasma sphingolipidome and phospholipidome in the metabolic syndrome. J Clin Endocrinol Metab. 2014 Nov;99(11):E2335-40. doi: 10.1210/jc.2014-1665. Epub 2014 Aug 20. PMID 25140396
- [Derived] Ooi EM, Watts GF, Chan DC, Chen MM, Nestel PJ, Sviridov D, Barrett PH. Dose-dependent effect of rosuvastatin on VLDL-apolipoprotein C-III kinetics in the metabolic syndrome. Diabetes Care. 2008 Aug;31(8):1656-61. doi: 10.2337/dc08-0358. Epub 2008 May 28. PMID 18509206
- [Derived] Ooi EM, Barrett PH, Chan DC, Nestel PJ, Watts GF. Dose-dependent effect of rosuvastatin on apolipoprotein B-100 kinetics in the metabolic syndrome. Atherosclerosis. 2008 Mar;197(1):139-46. doi: 10.1016/j.atherosclerosis.2007.03.004. Epub 2007 Apr 9. PMID 17416370